CLINICAL TRIAL: NCT01499680
Title: Multimodality Neuromonitoring In eXtreme Lateral Interbody Fusion (XLIF®)
Brief Title: Multimodality Neuromonitoring in XLIF
Acronym: NV in XLIF®
Status: Completed | Type: Observational
Sponsor: NuVasive (Industry)
Responsible Party: Sponsor
Organization: Globus Medical Inc (Industry)
Other Study IDs: NUVA.NV1001
Record Dates: First submitted 2011-12-02; First posted 2011-12-26 (Estimated); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Degeneration of Lumbar Intervertebral Disc
Keywords: Degenerative Lumbar Conditions

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- NV in XLIF: This group will have the XLIF procedure done using NV.

SUMMARY:
This is a prospective, non-randomized multi-center study to evaluate intraoperative neuromonitoring results in subjects who undergo eXtreme Lateral Interbody Fusion (XLIF) surgery at any number of levels inclusive of L4-5.

DETAILED DESCRIPTION:
Subjects will present with degenerative conditions in the lumbar spine that are amenable to surgical treatment and will be screened prior to study enrollment. Subjects will undergo neuromonitoring during the XLIF operation, as per standard care. They will then be re-evaluated immediately after surgery and at the first standard postoperative follow-up visit (6 weeks) to assess for presence of new neural deficit. If a new neural deficit is identified, the patient will be followed per the Investigator's standard follow-up schedule until symptoms have resolved (or are deemed permanent).

A total of 300 subjects will be enrolled in this study from multiple centers. The subjects will have degenerative conditions of the lumbar spine with planned treatment including XLIF surgery. The following eligibility criteria are designed to identify existing clinic patients for whom study under this protocol is considered appropriate. All subjects must meet the inclusion/exclusion criteria below in order to be considered for enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Persistent back and/or leg pain unresponsive to conservative treatment for at least six (6) months, unless surgical treatment is clinically indicated earlier
* Indicated for extreme lateral interbody fusion at any number of levels inclusive of L4-5
* At least 18 years of age at the date of written informed consent
* Able to undergo surgery based on physical exam, medical history and surgeon judgment
* Willing and able to return for post-treatment exams according to the follow-up called for in the protocol
* Signed and dated informed consent form

Exclusion Criteria:

* Patient has a mental or physical condition that would limit the ability to comply with study requirements
* Patient is a prisoner
* Patient is involved in active litigation relating to the spine (worker's compensation claim is allowed if it is not contested)
* Patient has an underlying neurological disease or neurological deficit that is not associated with the condition for which he/she is seeking surgical intervention (e.g., diabetic peripheral neuropathy)
* Patient is participating in another clinical study that would confound study data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population will consist of patients from participating site locations.
Sampling Method: Probability Sample
Enrollment: 323 (Actual)
Dates: Start 2011-10; Primary Completion 2013-12 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
The sensitivity and specificity of EMG and SSEP (if available) testing in identifying neural injury. | 8 weeks
  For evaluation of the primary endpoint and additional assessments, descriptive statistics including mean, standard deviation, minimum, median, and maximum for continuous variables and frequency distribution for categorical variables will be provided, as well as tabular listings. All complications will be itemized including incidence, duration, and relationship to devices used and/or procedures performed.

CONTACTS AND LOCATIONS:
Overall Officials: Kelli Howell, MS, Study Director — NuVasive
Locations (20):
- United States (18):
  - Shiley Center for Orthopaedic Research, La Jolla, California
  - UC Irvine Medical Center, Orange, California
  - Durango Orthopaedics, Durango, Colorado
  - USF Neurology and Neurosurgery, Tampa, Florida
  - West Augusta Spine Specialists, Augusta, Georgia
  - Georgia Spine and Neurosurgery Center, Decatur, Georgia
  - Pinnacle Orthopaedics and Sports Medicine, Marietta, Georgia
  - McLean Country Orthopedics, Bloomington, Illinois
  - Illinois Neurological Institute, Peoria, Illinois
  - Columbia Orthopaedic Group, Columbia, Missouri
  - Spine Midwest, Inc., Jefferson City, Missouri
  - Western Regional Center for Brain and Spine Surgery, Las Vegas, Nevada
  - Duke University Medical Center, Durham, North Carolina
  - South Oregon Spine Care, Medford, Oregon
  - Univerisity of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Coastal Orthopaedic Associates, Conway, South Carolina
  - Spine Pain Be Gone Clinic, San Antonio, Texas
- Caribbean Orthopaedic and Spine Institute, San Juan, PR, Puerto Rico
- Kantonsspital St. Gallen, Sankt Gallen, Switzerland